CLINICAL TRIAL: NCT05067686
Title: Health Professionals Perspective on Suicide: A Study of Their Attitude, Challenges and Suicide Prevention
Brief Title: Health Professionals Perspective on Suicide
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Syeda AYAT E ZAINAB Ali (Other)
Collaborators: University of Leicester (Other); University of Wuerzburg (Other)
Responsible Party: Sponsor-Investigator, Syeda AYAT E ZAINAB Ali, PhD Scholar, International Islamic University, Islamabad
Organization: International Islamic University, Islamabad (Other)
Other Study IDs: LWL-HPPS
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Suicide; Suicide, Attempted; Completed Suicide; Suicide Prevention
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicide, Completed; Suicide Prevention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mental Health Professionals
- Non Mental Health Professionals

SUMMARY:
The aim is to investigate how health professionals view/respond towards suicidal patients, what was their attitude, experiences and difficulties/challenges they faced while dealing with suicidal patients (whether successful or unsuccessful), and what measures/methods are optimal or could be used to prevent suicide from the perspective of mental and non mental health professionals through concurrent mixed methods study approach.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals having at least 1 year of experience in dealing with suicide cases irrespective of the outcome will be included.
* Qualification of Health professionals should be at least MBBS with permanent PMDCP registration.
* Health professionals who are willing to participate voluntarily and provide written informed consent will be included.

Exclusion Criteria:

* Health Professionals with prior and present history of psychiatric consultation will be excluded.
* Health Professionals without direct experience in handling suicidal patients will be excluded.
* Nurses and Paramedical staff will be excluded from the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Considering the study design (concurrent mixed methods), a sample size of sixteen health professionals from different specialties (n=4, Accident and Emergency, n=4 Medicine, n=4 Surgery, n=4 Mental Health) who are the front line clinicians dealing with suicidal behavior will be recruited for the qualitative study. For the quantitative study, the sample will comprised of ninety (n=100) health professionals from respective departments (n=50, (Non Mental Health Professionals, n=50 Mental Health Professionals). Data will be collected through purposive sampling technique.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03-29 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Interview Protocol for Qualitative Study | Day 1
  A interview protocol for qualitative study will comprised of detailed demographic sheet and open ended questions.

SECONDARY OUTCOMES:
The Understanding Suicidal Patients (USP) scale | Day 1
  The Understanding Suicidal Patients (USP) scale (Samuelsson, Asberg, & Gustavsson, 1997) will be used to measure willingness to provide care to suicide attempters and to assess the professional's understanding and sympathy for these patients.
The Stigma of Suicide Scale (SOSS-SF) | Day 1
  The Stigma of Suicide Scale (SOSS-SF) is a 16-item short form have been developed to examine attitudes towards "a prototypical person who completed suicide"
Attitudes towards Suicide Scale | Day 1
  The scale is used to examine the respondents' opinions and attitudes towards suicide. Factors measured by the scale are: (1) acceptability of suicide; (2) suicide as a sign of mental illness; (3) the belief that persons who commit suicide will be punished after death; (4) the opinion that suicidal people should communicate their problems; (5) the intention to hide past suicidal behavior; and (6) the opinion that suicide should be discussed and reported openly among friends or in the news.
Attitudes towards Suicide Prevention Scale | Day 1
  Attitude toward suicide prevention scale is a 14-item, self-rated, 5-point Likert scale (Strongly agree to strongly disagree) will be used to asses attitudes towards suicide prevention.
Difficulties in Suicidal Behaviors Intervention Questionnaire - Version for Psychologists and Doctors (DSBQ) | Day 1
  To assess the difficulties of health professionals when facing a patient who seeks help after a suicide attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tamkeen Saleem, PhD, Study Chair — International Islamic University, Islamabad, Pakistan; Dr Michelle O'Reilly, PhD, Study Chair — University of Leicester and Leicestershire Partnership NHS Trust; Dr Stefan M Schulz, PhD, Study Chair — University of Wuerzburg
Locations (1):
- International Islamic University, Islamabad Pakistan, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The impact of patient suicide on the professional reactions and practices of mental health caregivers and social workers — https://pubmed.ncbi.nlm.nih.gov/20801750/